CLINICAL TRIAL: NCT02582060
Title: Individualizing Hemophilia Prophylaxis Using Thromboelastography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Guy Young, Guy Young, MD, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-00030
Record Dates: First submitted 2015-10-09; First posted 2015-10-21 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Thrombelastography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Severe Hemophilia A Subjects (Other): The results of the TEG/ROTEM assay (specifically the R time/CT) will be used to determine the prophylaxis treatment regimen.
  Interventions: Other: Thromboelastography/Thromboelastometry-Guided Treatment Regimen

INTERVENTIONS:
Other: Thromboelastography/Thromboelastometry-Guided Treatment Regimen — The results of the TEG/ROTEM assay (specifically the R time/CT) will be used to determine the prophylaxis treatment regimen.

SUMMARY:
Currently dosing for prophylaxis is not individualized, and the general approach is to use a dose of 25-40 units/kg given 3 times per week or every other day. One of the issues with weight-based dosing is the possible over-treatment. This is likely due to the fact that laboratory tests are not sensitive enough at the low levels to support decision-making. The Thromboelastograph (TEG®) and Thromboelastometry (ROTEM®) are coagulation devices, which assess the dynamics of clot formation over time and have several characteristics which suggest they may provide important information for individualized prophylaxis treatment for our patients.

DETAILED DESCRIPTION:
This is a pilot study in children and adults with severe hemophilia A that utilizes the TEG/ROTEM to personalize their prophylaxis treatment.

Primary objectives:

• Assess the feasibility of TEG/ROTEM-guided modification of the current prophylaxis regimen for individuals with severe hemophilia A. Specifically, to:

* Test and refine the operational protocol for using TEG/ROTEM to guide factor dosing
* Estimate the proportion of hemophilia A patients whose dose will be modified based on TEG/ROTEM results
* Monitor short term safety of patients whose dose has been modified.

Secondary objectives

* Perform thrombin generation assays to provide additional evidence supporting the TEG/ROTEM-guided dosing.
* Obtain preliminary data on the economic impact of TEG/ROTEM-guided hemophilia A dosing regimens.
* Obtain preliminary data on the potential improvement of subject/family burden resulting from TEG/ROTEM-guided regimen using generic and specific quality of life tools.

The study period will consist of screening, pharmacokinetic (PK) study and follow-up. For subjects whose prophylaxis treatment regimen is modified, the follow-up period will include 3 follow-up clinic visits and 4 follow-up phone calls; these patients will remain on study for approximately 6 months following completion of the PK-study then will have an end of the study visit (visit 9). Subjects whose treatment regimen is not altered will end their study participation after Visit 2 and continuing with their current prophylaxis regimen.

Study endpoints: A safety review will be conducted after the first 6 subjects complete 30 days with the extended prophylaxis treatment. If no safety issues are identified, the study will proceed, and second safety review will be after an additional 8 subjects complete 30 days of extended treatment. If a subject has two or more spontaneous bleeds in 30 days, the subject will be removed from the study. For subjects who did not have bleeds and completed at least 6 months of the study, ongoing prophylactic treatment will be decided by their treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Males, 5-70 years, inclusive
* Plasma FVIII activity <1% documented (Laboratory result or MD documentation of Severe Hemophilia A diagnosis)
* Currently prescribed prophylaxis treatment regimen infusing ≥3 times a week
* Willing to alter their prophylaxis treatment regimen per study protocol

Exclusion Criteria:

* Bleeding disorder(s) other than Hemophilia A
* Current inhibitor (>0.6BU)
* Thrombocytopenia (platelet count <100,000K/µL since it can alter TEG®/ROTEM® results)
* Creatinine >2x the upper limit of normal (indicating potential platelet dysfunction)
* Prothrombin time >3 seconds above the upper limit of normal (indicating potential liver dysfunction)
* Any concurrent clinically significant major disease, frequent bleeding pattern or history of non-compliance that, in the opinion of the investigator, would make the subject unsuitable for enrollment
* Participation within the past 30 days in any other clinical study involving investigational drugs
* Planned major surgery within 30 days prior to screening or during the study period
* Current use of any medication known to have effects on the coagulation system

Ages: 5 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-05-20 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of TEG/ROTEM-guided prophylaxis modification for patients, assessed by estimated proportion of patients whose dose is modified. | Ongoing while patients are on study (~ 6 months)
  A total of 60 patients will be enrolled on this study. It is expected that less than 25% of these patients will be eligible for dose/schedule modification based on TEG/ROTEM.
Monitoring short-term safety of patients whose dose has been modified, assessed by monitoring number, type, and severity of bleeds. | Ongoing while patients are on study (~ 6 months)
  The primary endpoint for subject safety will be the occurrence of two serious spontaneous bleeding episodes within 28 days of each other.
Feasibility of TEG/ROTEM-guided prophylaxis modification for patients, assessed by testing and refining operational protocol for using TEG/ROTEM to guide factor dosing. | Ongoing while patients are on study (~ 6 months)

SECONDARY OUTCOMES:
Thrombin generation assay will be performed to provide additional evidence supporting the TEG/ROTEM-guided dosing. | 6 months
Assessment of direct costs for all subjects whose treatment was modified using factor consumption 6 months before, and the 6 months during study participation. | 1 year
  Analysis for those subjects who had a modified dosing regimen to determine the per capita reduction in consumption when a modified dosing regimen is achieved.
Assessment of indirect costs for all subjects whose treatment was modified using factor consumption 6 months before, and the 6 months during study participation. | 6 months
  Questionnaire collecting data on time spend on hemophilia-related care per week, caregiver support related to hemophilia, and number of infusions per week.
Improvement of subject/family burden as assessed by the Health-Related Quality of Life. | 6 months
  (HRQoL) Assessments/Analysis

CONTACTS AND LOCATIONS:
Locations (1):
- CHLA, Los Angeles, California, United States